CLINICAL TRIAL: NCT02786940
Title: Remote Cardiac Monitoring of Higher-Risk Emergency Department Syncope Patients After Discharge - A Pilot Study
Acronym: REMOSYNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 20160119-01H
Record Dates: First submitted 2016-03-21; First posted 2016-06-01 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Syncope; Arrhythmia
Keywords: remote; cardiac monitoring; mortality
MeSH Terms: conditions — Syncope; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Live Remote Cardiac Monitoring (Experimental): Patients in this arm will receive the Cardiophone device, a live remote cardiac monitoring with transmission of cardiac rhythm (device-triggered: if rhythm abnormalities detected by device algorithm; or patient-triggered by pressing the transmit button because of symptoms) for 15 days.
  Interventions: Device: Cardiophone
- Usual Care (Active Comparator): Patients in this arm will receive the Mobile Cardiac Telemetry device for 48-hour Holter monitoring as part of usual care. This device combines holter, event monitoring and mobile cardiac telemetry (continuous cardiac monitoring of every single beat) into one unit. The holter functionality will be used for the first 48 hours (usual care). The diagnostic yield from the 48 hour holter monitoring will be compared to the 15-day live monitoring.
  Interventions: Device: Cardiophone

INTERVENTIONS:
Device: Cardiophone — Remote live monitoring for 15 days for detection or exclusion of arrhythmias
  Other Names: ER920W event recorder, Braemar Inc

SUMMARY:
2-3% of emergency department (ED) syncope patients suffer arrhythmia/death within 30 days of disposition (either as an inpatient or at home) and we have recently developed the Canadian Syncope Risk Score (CSRS) to predict these outcomes. Currently, only Holter monitoring is used and is applied a few days later. New and innovative remote (out-of-hospital) external cardiac monitoring technology has made prolonged monitoring possible.

The primary objective is to compare diagnostic yield (identification of arrhythmia that requires treatment) for the following two strategies among higher-risk syncope patients discharged home from ED: 15-day external cardiac monitoring (intervention arm) versus 48-hour Holter monitor (control arm)

Methods: The study will be a double-blind RCT comparing two different approaches for detecting serious arrhythmias among high-risk ED syncope patients who are discharged home. Cardiophone (live monitor) will be used for the intervention arm and the Mobile Cardiac Telemetry (MCT) device will be used for the control arm and both devices applied prior to ED discharge. For patient safety purposes and to ensure that the patients are similar in both arms, all of the study patients will be monitored for 15 days. MCT will function as a holder for the first 48 hours and this will be used to compare the diagnostic yield in the two study arms. After written informed consent, patients will be randomized 1:1 with allocation concealed by web-based randomization and stratified based on the total CSRS scores.

Data collection: patient demographics, medical history, score predictors, device data (failure, false alarms, duration worn), patient symptoms, and comfort. The primary outcome will be the diagnostic yield at 15 days in the two study arms and primary analysis will compare the diagnostic yield by intention to treat principle controlling for the stratification factor. Sample Size: 300 patients per arm (600 total) to detect a 10% difference in diagnostic yield between the arms.

Impact: Our study will increase the early identification of patients with serious underlying arrhythmia by combining the CSRS risk tool with innovative remote monitoring technology.

DETAILED DESCRIPTION:
Syncope is a sudden transient loss of consciousness followed by spontaneous complete recovery; it is a very common problem and can be a precursor to sudden death. This study will increase the early identification of patients with serious underlying arrhythmia by combining our Canadian Syncope Risk Score (CSRS) with innovative remote (out-of-hospital) monitoring technology. Approximately 2-3% of ED syncope patients will suffer arrhythmia or die from unknown causes within 30 days of ED disposition (in-patient or outside the hospital). It is the concern for occult arrhythmia and its associated mortality that leads to prolonged cardiac monitoring in the ED, observation units, or by hospitalization; and wide variations in investigations and hospitalization. New and innovative technology has made remote monitoring feasible for prolonged periods (15-30 days) and is reliable. This technology allows arrhythmias to be transmitted live to a central monitoring station automatically based on the device algorithm or by the touch of a button when patients are symptomatic. However, the lack of tools to identify those at risk has limited the use of this new technology to improve patient outcomes. The CSRS tool, developed to predict the 30-day risk of arrhythmia/death showed that higher-risk (score ≥3) patients have a 17.2% observed risk of arrhythmia/death within 15 days. The aim of this randomized controlled trial (RCT) is to compare the diagnostic yield of a 15-day event monitor to a 48-hour Holter monitor (usual care) among higher-risk syncope patients discharged home at 10 Canadian EDs.

Context: Currently, only Holter monitoring (records all cardiac beats) for 1-2 days is used and prolonged monitoring devices are not used for arrhythmia detection. The majority of syncope patients are not monitored when symptomatic. Arrhythmias are detected only if evident when patients seek care. The investigators recently completed a multicenter prospective syncope study and developed the CSRS. Our results show that most serious conditions are identified within the first few hours in ED among low and moderate-risk patients while for non-low-risk patients the risk of arrhythmia remains high up to 15 days indicating the need for prolonged monitoring.

Previous studies and Rationale: A small randomized study with the old technology that required patient activation for arrhythmia capture found higher diagnostic yield than Holter, but the utility was limited due to patients' inability to activate the device after symptoms. Two small studies of unselected syncope patients, one prospective (n=48) and another registry analysis (n=92) found a diagnostic yield of 30 - 38% with prolonged monitoring for 7-33 days. The diagnostic yield of Holter is 1-20% based on the risk of enrolled patients. The role of prolonged cardiac monitoring among ED syncope patients has not been well studied. Only Holter monitoring is being currently used, but inconsistently and is applied a few days later. With the technological advances, the investigators hypothesize that 15-day monitoring will lead to higher diagnostic yield than Holter and plan to apply the devices before disposition for high-risk patients discharged home.

Objectives: The primary objective of the REMOSYNC study is to compare diagnostic yield (identification of arrhythmia that requires treatment or exclusion of an arrhythmic cause) for the following two strategies in higher-risk ED syncope patients discharged home from ED: 15-day external cardiac event monitoring (intervention arm) versus 48-hour Holter monitoring (control arm).

Design and Setting: The study will be a multicenter two-arm, double-blinded randomized controlled trial (RCT) comparing two different approaches for detecting serious arrhythmias among high-risk ED syncope patients who are discharged home. Half of the study patients will be randomized to 15-day external cardiac monitoring (intervention group) and the other half will be assigned to 48-hour Holter monitoring (control group and current practice pattern).

Patient Recruitment: Consecutive patients who fulfill inclusion and do not meet any exclusion criteria will be approached for recruitment at the participating EDs and enrolled after informed written consent.

Randomization: Patients will be randomized in a 1:1 ratio to either receive a 15-day event monitor Cardiophone (intervention arm) or a 48-hour Holter monitoring with the MCT device (control arm). Patients will be stratified based on the total CSARS score: 3-4; 5-6; and 7-8 and allocated using randomly permuted blocks of varying lengths. Allocations will be computer-generated by an independent statistician and concealed by having research staff log on to a password-protected Electronic Data Capture (EDC) System located within the coordinating center website.

Intervention: Enrolled patients will receive all outpatient investigations except monitoring (which will according to the randomization as per the study protocol) as per the discharging physician. Based on their allocation, patients will receive either Cardiophone or the MCT device prior to discharge home. The allocation will be concealed and the treating physician, patient, outcome assessor, and the investigator will be blinded to the arm the patient is randomized.

Data Collection: Patient demographics, medical history, CSRS predictors, results of physical examination and investigations, and patient disposition will be collected. The following device data will be obtained from the central monitoring station: quality of recordings, device failure (rhythm not captured during death or when symptomatic), false alarms due to artifacts, times of patient activation of cardiophone device due to symptoms, any rhythm abnormalities detected during the symptoms, and monitoring reports for patients in both arms. Patients will complete a questionnaire during the follow-up visit regarding any serious conditions suffered, their comfort, and how secure they felt because of the cardiac monitoring.

Post-ED Care of Study Patients: All patients enrolled in the study will be linked to a local cardiology group for any urgent and end-of-study follow-up as needed. Patients will be advised to keep a diary of symptoms during the 15-day monitoring period. Patients in the cardiophone arm will have the option of transmitting the rhythm when symptomatic and symptom-rhythm correlation will be reported. Patients will be advised to return the devices and the symptom diary to the local cardiology clinic or the ED research team the next business day after the 15-day monitoring period. All monitoring reports will be completed by the central monitoring station within 24 hours and sent to the study cardiologist. If serious arrhythmias are detected, then the central monitoring station will contact the patient or the family member and advise them to call 911 for the patient to be transported to the ED. If other arrhythmias are identified, the central monitoring station will provide an interim report to the study cardiologist providing care. The study cardiologist will decide the need for urgent follow-up and the time frame within which such follow-up should occur. For patients in the control arm with an MCT device, the central monitoring station will provide reports for 48-hour Holter monitoring on day 3 and another report on day 16 for cardiac monitoring for days 3 to 15. Patients in both study arms will be clearly advised to seek care for symptoms as usual. All patients will be monitored for the entire 15 days regardless of early arrhythmias detected and will have end-of-study follow-up and further management as deemed appropriate by the cardiologist responsible for the care of the patient.

Duration of Participation and Withdrawal: Patients will be part of the study actively for 1-year after recruitment. We plan to conduct a 30-day telephone follow-up and 1-year health administrative data linkage for serious outcomes related to syncope. Patients will be free to withdraw from the study at any time without providing any reason and without any penalty or loss of benefits they are entitled and the number of withdrawals will be monitored. However, as these monitoring devices will serve to allay the fear of arrhythmia or death among patients, the investigators expect very few withdrawals. There will be no restrictions on medications or procedures during the study period.

Data Analysis: The primary analysis will be by intent-to-treat and will compare the diagnostic yield (arrhythmia detection or exclusion) at the end of 15 days using data from 15-day monitoring in the intervention arm and the 48-hour Holter monitoring. The secondary analysis will include a per-protocol analysis. The Cochran-Mantel-Haenszel test will be used for the primary outcome, controlling for the stratification factor (CSRS score). The effect of the intervention will be expressed as a risk difference with 95% confidence interval. Secondary analysis will include multivariable logistic regression to control for potential confounders or imbalances between patients in the study arms. Descriptive statistics for baseline characteristics, all outcomes, device performance including failure, and patient-centered measures (adherence, comfort, and safety feeling). Additional analysis will include a comparison of arrhythmias detected that did not require treatment between the groups. There will be no interim analyses for efficacy performed, but the investigators will monitor trial safety as detailed in the Data Safety Monitoring Board section.

Sample Size: Our sample size is 300 patients per arm (600 total) determined to yield 80% power to detect an absolute difference of 10% in diagnostic yield between the study arms using a chi-squared test at the 5% level of significance assuming a control arm event rate of 17% and accounting for 5% attrition. A difference of 10% is feasible based on previous studies which have reported an 18% increase in diagnostic yield with prolonged monitoring.

Data Safety Monitoring Board: This independent committee will be comprised of one emergency physician, one cardiologist, and a biostatistician from outside the participating sites. This board will be responsible for safeguarding the interests and safety of trial participants by reviewing adverse events including deaths every 6 months during the study period.

Anticipated Contributions: Our study will be the first to combine risk stratification and innovative technology to decrease morbidity and mortality, and improve healthcare efficiency. This study will create new knowledge regarding the role of prolonged live monitoring among high-risk syncope patients and the application of devices prior to ED discharge. As the monitoring is live, timely management of potentially life-threatening arrhythmias is possible and can be applied to syncope patients, not at risk for ventricular arrhythmia and hospitalized solely for cardiac monitoring. This will represent a paradigm shift as patients can now be monitored at home at a very low cost decreasing ED and hospital crowding. These devices will alleviate fears of occult arrhythmia and death and will improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age ≥18 years) patients with syncope
2. High-risk as per the Canadian Syncope Risk Score (score > or =3)and being discharged home after ED physician or consultant assessment.

Exclusion Criteria:

1. Syncope patients with a score <3
2. Those who are hospitalized
3. Previously enrolled.
4. Loss of consciousness not related to syncope: prolonged loss of consciousness > 5 minutes
5. Change in the mental status from baseline
6. Patients with alcohol intoxication or illicit drug abuse, witnessed obvious seizure; or head trauma, i.e. trauma the initial event.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Proportion of participants among whom arrhythmias are detected that required treatment | 15-days
  The primary outcome will be the diagnostic yield and includes detection of serious arrhythmias that required treatment or that caused death. The investigators will collect data on the type of treatment offered (medications; implantable loop recorder, pacemaker, defibrillator, or dual device insertions; cardioversion or therapeutic ablation). A blinded Adjudication Committee of 3 physicians will confirm all outcomes.

SECONDARY OUTCOMES:
Exclusion of arrhythmia | 15-days
  Secondary outcomes include arrhythmias for which treatment was not offered. Treatment for arrhythmias include medications, implanatation of pacemaker, defibrillator, or dual device; cardioversion or therapeutic ablation). A blinded Adjudication Committee of 3 physicians will confirm that the arrhythmia identified did not require the above treatments.
  If a normal sinus rhythm was identified at the time of syncope, then we will report that no arrhythmia was identified during the syncope
Detection of arrhythmias that did not require treatment | 15 days
  Secondary outcomes include arrhythmias for which treatment was not offered. Treatment for arrhythmias include medications, implanatation of pacemaker, defibrillator, or dual device; cardioversion or therapeutic ablation). A blinded Adjudication Committee of 3 physicians will confirm that the arrhythmia identified did not require the above treatments.
  If a normal sinus rhythm was identified at the time of syncope, then we will report that no arrhythmia was identified during the syncope
Safety of the live monitoring device | 15 days
  The investigators will report the proportion of patients with adverse events due to device failure.
  In both arms:
  1. The duration of time the devices were worn will be reported.
  2. The proportion of patients with arrhythmias that did not require treatment will be reported.
Compliance of the participants in wearing the devices | 15 days
  The duration the devices were worn will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Thiruganasambandamoorthy, MBBS, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No